CLINICAL TRIAL: NCT07121491
Title: The Effect Of Zhang's Guidelines Versus Who Partograph On Childbirth Experience According To Ceq-My
Brief Title: Effects and Childbirth Experience Between Zhang and WHO Partograph
Status: Completed | Type: Observational
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Rahana Abd Rahman, Associate Professor, National University of Malaysia
Other Study IDs: FF-2024-280
Record Dates: First submitted 2025-07-24; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Outcome, Adverse Birth; Childbirth Experience
Keywords: Labour outcome; Childbirth experience
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cervical dilatation 4 cm: Women with cervical dilatation 4 cm
- Cervical dilatation 6 cm: Women with cervical dilatation 6 cm

SUMMARY:
This study compared the labour outcomes and childbirth experience between Zhang and WHO partograph.

DETAILED DESCRIPTION:
A prospective cross-sectional observational study that compared the cervical os dilatation i.e 4 and 6 cm upon admission to the labour room. Eligible patients were recruited during postnatal period in the ward before discharged home. The details of clinical characteristics and labour outcomes were collected. Patients then answered the CEQ-My questionnaire form that assess their childbirth experiences. The primary outcome measure was caesarean section rate and the secondary outcome measure was the childbirth experience.

ELIGIBILITY:
Inclusion Criteria:

* cervical dilatation 4 or 6 cm
* singleton
* cephalic presentation
* at 37 weeks or more
* normal cardiotocograph tracing on admission
* understands Malay or English
* no uterine scar
* no pre-existing medical disorders
* no antenatal complications such as diabetes or hypertension

Exclusion Criteria:

* multiple pregnancy
* none cephalic presentation
* abnormal admission cardiotocograph tracing
* less than 37 weeks gestation
* refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women genetically XX
Study Population: All women who fulfil the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 713 (Actual)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Caesarean section rate | from cervical dilatation of 4 or 6 cm through study completion up to delivery of the foetus
  Rate of delivery via caesarean section in percentage

SECONDARY OUTCOMES:
Childbirth experience | from Day 1 throughout study completion, an average of 7 days after delivery
  Assessment of experience during delivery using questionnaire based on based on total childbirth experience questionnaire score using Likert scale from 1 to 4. Score of 4 is a total agreement and score of 1 is total disagreement.

OTHER OUTCOMES:
Use of analgesia | From cervical dilatation of 4 or 6 cm until delivery of fetus
  Number of patients needed analgesia in percentage
Oxytocin use | From cervical dilatation of 4 or 6 cm until delivery of fetus
  Number of women who needed oxytocin infusion
Duration of hospital stay | From predelivery throughout study completion, an average of 5 days
  Duration from admission until discharge either 3 days or less or more than 3 days
Admission into neonatal care intensive unit | From birth of the neonate until throughout study completion, an average of 7 days after birth
  Number of neonates needed to be admitted into neonatal care intensive unit
Apgar score at 5 minutes | From delivery of neonate until 5 minutes after delivery
  Neonatal Apgar score less than 7 at 5 minutes after delivery based on the Apgar score with 0 the lowest and 10 the highest

CONTACTS AND LOCATIONS:
Overall Officials: Rahana Abd Rahman, Principal Investigator — National University of Malaysia
Locations (1):
- Hospital Canselor Tuanku Muhriz, Kuala Lumpur, Cheras, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon request